CLINICAL TRIAL: NCT03638089
Title: Fall Recovery Training for Individuals With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Jeremy Crenshaw, Assistant Professor, University of Delaware
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 791562-8
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): This group will receive up to six sessions of fall-recovery training over the course of 2-3 weeks.
  Interventions: Behavioral: Fall-recovery training

INTERVENTIONS:
Behavioral: Fall-recovery training — Participants practice recovering from simulated, treadmill-induced slips and trips.

SUMMARY:
The purpose of this study is to quantify how fall-recovery training improves the fall-recovery response of individuals with chronic stroke. Up to 20 participants with chronic stroke will be recruited from the community. Over six laboratory visits, participants will undergo sessions of fall-recovery training. Each session is comprised of simulated trips and slips as participants stand on a computer-controlled treadmill. Trip-recovery training consists of treadmill-delivered disturbances that induce a forward fall. Slip-recovery training consists of a treadmill-delivered disturbances that induce a backward fall. Separate progressions focus on initial steps with the left and right limbs. The training intensity, as determined by the disturbance magnitude, is progressive and dependent on participant performance. Step length and maximum trunk angle will be calculated. The hypothesis is that, with practice, participants will recover from larger perturbations, and they will increase step length and reduce trunk rotation during fall recoveries.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older
* Participants must have had a single stroke of non-cerebellar origin

Exclusion Criteria:

* More than one stroke
* Unable to walk one block without stopping or using a walking aid, such as a cane
* Acute illness at the time of functional assessment or training
* Body mass greater than 136 kg (300 lbs)
* Lower extremity joint replacement or shoulder joint replacement within a year prior to participation
* Dementia
* Parkinson's disease
* A history of back surgery
* A history of neck surgery
* More than one occurrence of back or neck pain in the month prior to participation
* Current back or neck pain at the time of participant enrollment
* Bulging vertebral discs
* Spine, hip, or lower extremity fracture within a year prior to participation
* Open lesions on the lower extremity
* Insulin-dependent diabetes
* Use of a pacemaker
* Use of an ostomy pouch
* Pregnancy
* Osteoporosis
* Doctor recommendation to avoid moderate physical activity or exercise
* Any neural, muscular, or skeletal condition or injury that precludes safe participation in the training or introduces a confounding factor on the study, at the discretion of the clinician or study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Disturbance magnitude | 2-3 weeks (first to last training session)
  The highest disturbance magnitude from which a successful fall-recovery resulted on the first and last training sessions

SECONDARY OUTCOMES:
Step length | 2-3 weeks (first to last training session)
  The length of the initial recovery step in response to the highest disturbance magnitude common to the first and last training sessions
Trunk rotation | 2-3 weeks (first to last training session)
  The maximum trunk rotation angle in response to the highest disturbance magnitude common to the first and last training sessions

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pigman J, Reisman DS, Pohlig RT, Wright TR, Crenshaw JR. The development and feasibility of treadmill-induced fall recovery training applied to individuals with chronic stroke. BMC Neurol. 2019 May 25;19(1):102. doi: 10.1186/s12883-019-1320-8. PMID 31128598